CLINICAL TRIAL: NCT04668651
Title: Preoperative Evaluation of Gastric Contents by Antral Ultrasound in Diabetic Patients: a Prospective Observational Study
Brief Title: Preoperative Evaluation of Gastric Contents by Antral Ultrasound in Diabetic Patients
Acronym: PEGASED
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator has left Nice University Hospital and no other doctor has taken over for the study.
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20-PP-17
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic: diabetic patients
  Interventions: Other: antral ultrasound
- non diabetic: non-diabetic patients
  Interventions: Other: antral ultrasound

INTERVENTIONS:
Other: antral ultrasound — Preoperative evaluation of gastric contents by antral ultrasound

SUMMARY:
Gastric aspiration represents the third cause of perioperative death in France. In scheduled surgery, it can be prevented by preoperative fasting. The French and American guidelines recommend a fasting of 2 hours for clear liquids and 6 hours for solid food. However, these durations could be too short in case of delayed gastric emptying due to medications of diabetes for example. This latter condition has an increasing incidence. Numerous complications are related to chronic hyperglycemia including delayed gastric emptying also known as gastroparesis. Around one third of diabetic patients presents this complication.

Gastric ultrasound represents a non-invasive method to explore the stomach. It allows the qualitative and quantitative evaluations of gastric content.

As diabetic patients present a risk of non-empty stomach despite fasting,investigators decided to conduct a prospective observational study compare the appearance of the stomach assessed by ultrasonography between diabetic and non-diabetic patients before scheduled surgery

DETAILED DESCRIPTION:
Gastric aspiration represents the third cause of perioperative death in France. The physiopathology of this complication is multifactorial, implying among other things the lack of respect for the rules of preoperative fasting, especially during emergency operations. Indeed, the presence of food content in the stomach, combined with the decrease in the pressure of the lower sphincter of the esophagus and the protection of the upper airways during the induction of general anesthesia, is accompanied by a significant increase in the risk of regurgitation and inhalation of gastric contents.

There are more than 3 million diabetic patients in France, with an increase in prevalence of more than 5% per year. The main digestive disorder linked to autonomic neuropathy in the diabetic subject is represented by gastroparesis, characterized by a delay in gastric emptying without mechanical impediment, associated with signs of abnormal gastric motility. Gastroparesis results from an impairment of the neurovegetative regulation of the stomach related to exposure to prolonged hyperglycemia. It is estimated that approximately 1/3 of diabetics are affected.

Ultrasound measurement of the antral section area was originally described for the evaluation and study of gastric emptying in obstetrics and medicine. Several studies have shown the interest of this measurement for the evaluation of gastric content and volume in the preoperative period. The antral ultrasound makes it possible to discriminate a "full" stomach from an "empty" stomach with excellent performance. Thus, investigators have at our disposal a simple and non-invasive tool to evaluate in real time the state of gastric vacuity in patients in the operating room.

In practice, ultrasound measurement of the antral section area is performed using an ultrasound scanner equipped with a 2-5 MHz frequency probe. The diameters (longitudinal D1 and anteroposterior D2) of the antrum are measured in the sagittal plane passing through the abdominal aorta and the left lobe of the liver. The value of the antral cross-sectional area is given by the formula: antral area = π x D1 x D2 / 4. This ultrasound measurement of the antral cross-sectional area is commonly performed in the operating room and is recommended in some anesthesia reference books. Several mathematical models have been constructed, in adults and children, to calculate the volume of gastric contents based on this measurement of anal area, with satisfactory accuracy (R² = 0.72 to 0.86). Gastric ultrasound is easily performed at the patient's bedside, before general or local anesthesia, and its use has recently been described to study gastric emptying.

Investigators would like to evaluate the gastric content in diabetics in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Any treated diabetic and non-diabetic patient requiring elective vascular surgery who has agreed to participate in the study (consent form obtained).
* Affiliation or beneficiary of social security.

Exclusion Criteria:

* Pregnant woman
* Persons of full age protected by law
* Patient Refusal
* Patient deprived of liberty
* History of gastric surgery
* Any situation requiring urgent treatment that is not compatible with the performance of a gastric ultrasound scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any treated diabetic and non-diabetic patient requiring elective vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Antral content | Preoperative
  Evaluation of antral content according to the Perlas classification (0, 1 or 2) and antral surface area between diabetic and non-diabetic patients.

SECONDARY OUTCOMES:
Antral area | Pre-operative, on arrival in the operating room
  Evaluation of antral surface area between diabetic and non-diabetic patients
Perlas grades | Pre-operative, on arrival in the operating room
  Evaluation of Perlas grades between diabetic and non-diabetic patients
Characteristics of diabetes | Pre-operative, on arrival in the operating room
  Correlate the antral surface area and characteristics of diabetes (type, duration, glycosylated hemoglobin results)
Clinical signs of diabetic gastroparesis | Pre-Anesthesia Consultation
  Evaluation of antral surface area and clinical signs of diabetic gastroparesis
Perioperative respiratory complications | Peri-operative
  Correlate the antral surface and perioperative respiratory complications: inhalation, pneumopathy and respiratory distress

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ORBAN, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, PACA, France